CLINICAL TRIAL: NCT05060263
Title: A Phase 1, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of HOT1030 in Patients With Advanced Solid Tumors
Brief Title: A Study of of HOT1030 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HOT-1030-1
Record Dates: First submitted 2021-03-26; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Intervention Model Description: dose-escalation study
Masking Description: open-label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): HOT-1030, every 21 days by intravenous administration. HOT-1030 is a recombinant humanized CD137 monoclonal antibody injection.
  Interventions: Drug: HOT-1030
- Cohort 2 (Experimental): HOT-1030, every 21 days by intravenous administration. HOT-1030 is a recombinant humanized CD137 monoclonal antibody injection.
  Interventions: Drug: HOT-1030
- Cohort 3 (Experimental): HOT-1030, every 21 days by intravenous administration. HOT-1030 is a recombinant humanized CD137 monoclonal antibody injection.
  Interventions: Drug: HOT-1030
- Cohort 4 (Experimental): HOT-1030, every 21 days by intravenous administration. HOT-1030 is a recombinant humanized CD137 monoclonal antibody injection.
  Interventions: Drug: HOT-1030
- Cohort 5 (Experimental): HOT-1030, every 21 days by intravenous administration. HOT-1030 is a recombinant humanized CD137 monoclonal antibody injection.
  Interventions: Drug: HOT-1030
- Cohort 6 (Experimental): HOT-1030, every 21 days by intravenous administration. HOT-1030 is a recombinant humanized CD137 monoclonal antibody injection.
  Interventions: Drug: HOT-1030
- Cohort 7 (Experimental): HOT-1030, every 21 days by intravenous administration. HOT-1030 is a recombinant humanized CD137 monoclonal antibody injection.
  Interventions: Drug: HOT-1030

INTERVENTIONS:
Drug: HOT-1030 — HOT-1030 is a Recombinant Humanized CD137 Monoclonal Antibody Injection
  Other Names: no other interventions

SUMMARY:
A Phase 1, Open-label, Dose-escalation Study of the Safety and Pharmacokinetics of HOT-1030 in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
This study is an open-label, Phase 1, study to evaluate the safety, tolerability, PK, and PD profiles of HOT-1030 as a monotherapy to assess the maximum tolerated dose (MTD) in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female from 18 to 75 yrs (include 18 yrs and 75 yrs).
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
3. Patients with histologically or cytologically confirmed advanced malignant solid tumor who have received or been intolerant of all standard therapies thought to confer clinical benefit.
4. Measurable disease on imaging base on RECIST v1.1 for solid tumors;
5. Stop anticancer therapy for more than 5 half-lives or 4 weeks (whichever is shorter) prior to study entry;
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
7. Adequate organ function, as indicated by the laboratory values.
8. Female patients of childbearing potential must have a negative serum pregnancy test at screening; Male patients and the female patients of childbearing potential must agree to use highly effective contraceptive measures throughout the study starting with the Screening Visit through 90 days after the last dose of study treatment is received.
9. Life expectancy >3 months.

Exclusion Criteria:

1. Received any anti-CD137 antibodies.
2. Active primary CNS tumor or metastatic CNS tumor (expect the patients who had received the treatment and stopped the treatment for more than 4 weeks before first dose), active epilepsy, Spinal cord compression or Cancerous meningitis.
3. Active autoimmune disease or history of autoimmune disease requiring systemic therapy < 2 years prior to screening except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes. Patients with childhood asthma or atopy that has not been active in the 2 years prior to study screening are eligible.
4. Require systematic anti-infective therapy a week before first dose because of active infection.
5. Taken the surgical operations not related to the research 4 weeks before first dose
6. Used of systemic corticosteroids (a dose equivalent > 10 mg/day of prednisone or )or other immunosuppressive agents, excepted:

   1. Patients are allowed to have topical use or inhaled glucocorticoid.
   2. Patients are allowed to have a less than seven-day glucocorticoid treatment preventing or treat non-autoimmune allergic diseases.
7. The toxicity of previous anti-tumor therapy has not recovered (defined as not recovering to grade 0 or 1, except for alopecia) or has not fully recovered from previous surgery.
8. During the 6 months prior to screening, the patient had a history of major cardiovascular and cerebrovascular events, such as myocardial infarction, coronary angioplasty or bypass surgery, heart valve repair, unstable arrhythmias, unstable angina, transient ischemic attack, or cerebrovascular accidents.
9. New York Heart Association (NYHA) grade III or IV congestive heart failure.
10. Patients with uncontrolled hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥100mmHg at the time of screening) who had been on a stable dose of antihypertensive drugs for at least 4 weeks at the time of screening).
11. Active hepatitis B (hepatitis B virus titer >103 copies /ml or 200IU/ml); Hepatitis C virus infection (HCV-RNA above the detection limit); Prophylaxis antiviral therapy other than interferon is allowed. In patients with advanced liver cancer (HCC), hepatitis B virus titer >104 copies /ml or 2000IU/ml should be excluded.
12. A history of known congenital and acquired immunodeficiency, including positive HIV antibody tests.
13. Patients with a known history of severe allergic reactions to macromolecular protein formulations/monoclonal antibodies or to any investigational drug component (CTCAE V5.0 grade greater than 3).
14. Participated in clinical trials of other drugs within 4 weeks before the first administration.
15. Pregnant or lactating women or women at risk of pregnancy have a positive pregnancy test before the first medication.
16. Other investigators consider that the patient has any clinical or laboratory abnormality that makes him unsuitable for participation in this clinical study.
17. prior history of a clear neurological or psychiatric disorder, including epilepsy or dementia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as measured by incidence of AEs (Adverse Events) | through study completion， an average of 1 year
  Incidence and severity of AEs, Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

SECONDARY OUTCOMES:
Area Under Curve (AUC) of HOT-1030 | 42 days
  Area under the concentration-time curve of HOT-1030 in plasma over the time interval from 0 extrapolated to infinity
Maximum Serum Concentration (Cmax) of HOT-1030 | 42 days
  Maximum Serum Concentration (Cmax) in plasma
Antitumor Activity of HOT-1030 in Patients With advanced Solid Tumors | through study completion， an average of 1 year
  Response is defined as a Complete Response + Partial Response and was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Han Baohui, Doctor, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Huaota Biopharmaceutical Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No